CLINICAL TRIAL: NCT00351468
Title: EXTEND (Eltrombopag Extended Dosing Study): An Extension Study of Eltrombopag Olamine (SB-497115-GR) in Adults, With Idiopathic Thrombocytopenic Purpura (ITP), Previously Enrolled in an Eltrombopag Study.
Brief Title: EXTEND (Eltrombopag Extended Dosing Study)
Acronym: EXTEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRA105325
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: eltrombopag olamine; SB-497115-GR; idiopathic thrombocytopenic purpura; thrombocytopenia; ITP; platelets
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag (Experimental): Open-label eltrombopag
  Interventions: Drug: eltrombopag olamine (SB-497115-GR)

INTERVENTIONS:
Drug: eltrombopag olamine (SB-497115-GR) — Eltrombopag with starting dose of 50mg daily, max dose of 75mg daily and min dose of 25mg daily or less frequently. Modifications were given to maintain platelet count in range of 50 to 200 Gi/L.

SUMMARY:
An open-label, dose-adjustment, extension study to evaluate the safety and efficacy of eltrombopag for the treatment of subjects with idiopathic thrombocytopenic purpura (ITP) who have previously been enrolled in an eltrombopag trial. This study will allow adjustment of the eltrombopag dose to achieve an individualized dose and schedule for each subject. In addition, the ability to reduce the dose of concomitant ITP medications in the presence of eltrombopag, while maintaining platelet counts = 50,000/μL will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated a written informed consent.
* Adults (≥18 years) diagnosed with ITP according to the American Society for Hematology/British Committee for Standards in Haematology (ASH/BCSH) guidelines [George, 1996; BCSH, 2003]. In addition, a peripheral blood smear should support the diagnosis of ITP with no evidence of other disease causative of thrombocytopenia (e.g., pseudo thrombocytopenia, myelofibrosis). The physical examination should not suggest any disease which may cause thrombocytopenia other than ITP.
* Prior completion of treatment and follow up periods in an ITP study of eltrombopag (e.g., TRA100773 or TRA102537/RAISE or TRA108057/REPEAT).
* Subjects previously enrolled in Study TRA100773 must have completed the prescribed follow-up ophthalmic assessment at 6 months.
* Subjects previously enrolled in TRA102537/RAISE or other studies that may lead into EXTEND (e.g., TRA108057/REPEAT) must have completed the treatment and follow-up periods as defined in that protocol.
* Subject experienced no eltrombopag-related toxicity or other drug intolerance on prior eltrombopag study (e.g., TRA100773 or TRA102537/RAISE or TRA108057/REPEAT) even if resolved; subjects discontinued from previous study due to toxicity will not be eligible unless they received placebo.
* Subject has no intercurrent medical event, including thrombosis.
* Subjects must have either initially responded (platelet count > 100,000/mL) to a previous ITP therapy or have had a bone marrow examination consistent with ITP within 3 years to rule out myelodysplastic syndromes or other causes of thrombocytopenia
* Previous therapy for ITP with immunoglobulins (IVIg and anti-D) must have been completed at least 1 week prior to first dose of study medication and the platelet count must show a clear downward trend after the last treatment with immunoglobulins. Previous treatment for ITP with splenectomy, rituximab and cyclophosphamide must have been completed at least 4 weeks prior to randomization, or clearly be ineffective.
* Subjects treated with concomitant ITP medication (e.g. corticosteroids or azathioprine) must be receiving a dose that has been stable for at least 4 weeks prior to randomization. Subjects treated with cyclosporine A, mycophenolate mofetil or danazol must be receiving a dose that has been stable for at least 3 months prior to the first dose of study medication.
* Prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) must be within 80 to 120% of the normal range with no history of hypercoagulable state.
* A complete blood count (CBC), within the reference range (including WBC differential not indicative of a disorder other than ITP), with the following exceptions:
* Hemoglobin: Subjects with hemoglobin levels between 10.0 g/dL and the lower limit of normal are eligible for inclusion, if anemia is clearly attributable to ITP (excessive blood loss).
* ANC≥1500/mL (1.5 x 10^9/L) is required for inclusion (elevated WBC/ANC due to steroid treatment is acceptable).
* The following clinical chemistries MUST NOT exceed the upper limit of normal (ULN) reference range by more than 20%: creatinine, ALT, AST, total bilirubin, and alkaline phosphatase. In addition, total albumin must not be below the lower limit of normal (LLN) by more than 10%.
* Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use one of the following highly effective methods of contraception (i.e., Pearl Index <1.0%) from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:
* Complete abstinence from intercourse;
* Intrauterine device (IUD);
* Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide);
* Male partner is sterile prior to entry into the study and is the only partner of the female;
* Systemic contraceptives (combined or progesterone only).
* Subject is able to understand and comply with protocol requirements and instructions.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Any clinically relevant abnormality, other than ITP, identified on the screening examination, or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another diagnosis.
* Concurrent malignant disease and/or history of cancer treatment with cytotoxic chemotherapy and/or radiotherapy.
* Any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), AND≥two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, etc), or any other family history of arterial or venous thrombosis
* Pre-existing cardiovascular disease (including congestive heart failure, New York Heart Association [NYHA] Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec.
* Female subjects who are nursing or pregnant (positive serum or urine b-human chorionic gonadotrophin (b-hCG) pregnancy test) at screening or pre-dose on Day 1.
* History of alcohol/drug abuse.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* Subject treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDs) or anti-coagulants for > 3 consecutive days within 2 weeks of the study start and until the end of the study.
* History of platelet agglutination abnormality that prevents reliable measurement of platelet counts.
* All subjects with secondary immune thrombocytopenia, including those with laboratory or clinical evidence of HIV infection, antiphospholipid antibody syndrome, chronic hepatitis B infection, hepatitis C virus infection, or any evidence for active hepatitis at the time of subject screening. If a potential subject has no clinical history that would support HIV infection or hepatitis infection, no further laboratory screening is necessary; however, standard medical practice would suggest further evaluation of patients who have risk factors for these infections.
* A subject is planning to have cataract surgery.
* In France, a subject is neither affiliated with nor a beneficiary of a social security category.

Other Eligibility Criteria Considerations:

To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the following document(s) for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the investigational product(s) being used in this study: CIB, SPM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2006-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (103):
- United States (23):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Brunsville, Minnesota
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, Arlington, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Vancouver, Washington
- Australia (2):
  - Novartis investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Kogarah, New South Wales
- Novartis Investigative Site, Vienna, Austria
- Canada (2):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (3):
  - Novartis Investigative Site, Jiang Su Province
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Odense, Denmark
- Novartis Investigative Site, Kuopio, Finland
- France (3):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Pessac
- Germany (5):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Giessen, Hesse
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Saarbrücken, Saarland
  - Novartis Investigative Site, Berlin, State of Berlin
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Shatin, New Territories, Hong Kong
- Italy (4):
  - Novartis Investigative Site, Bologna, Emilia-Romagna
  - Novartis Investigative Site, Albano Laziale (Roma), Lazio
  - Novartis investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Padua, Veneto
- Netherlands (5):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, The Hague
- New Zealand (4):
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Grafton
  - Novartis Investigative Site, Takapuna, Auckland
- Pakistan (2):
  - Novartis Investigative Site, Karachi
  - Novartis Investigative Site, Lahore
- Peru (2):
  - Novartis Investigative Site, Lima, Lima Province
  - Novartis Investigative Site, Lima
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Bucharest, Romania
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis investigative Site, Saint Petersburg
- Slovakia (2):
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Prešov
- Novartis Investigative Site, Ljubljana, Slovenia
- Novartis Investigative Site, Seoul, South Korea
- Spain (6):
  - Novartis Investigative Site, Badalona/Barcelona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Santiago de Compostela
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Novartis Investigative Site, Taipei, Taiwan
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Khon Kaen
- Tunisia (4):
  - Novartis investigative Site, Montfleury
  - Novartis investigative Site, Sfax
  - Novartis Investigative Site, Sousse
  - Novartis Investigative Site, Tunis
- Ukraine (2):
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Lviv
- United Kingdom (7):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Reading
  - Novartis Investigative Site, Swansea
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Wong RSM, Saleh MN, Khelif A, Salama A, Portella MSO, Burgess P, Bussel JB. Safety and efficacy of long-term treatment of chronic/persistent ITP with eltrombopag: final results of the EXTEND study. Blood. 2017 Dec 7;130(23):2527-2536. doi: 10.1182/blood-2017-04-748707. Epub 2017 Oct 17. PMID 29042367
- [Derived] Tarantino MD, Fogarty P, Mayer B, Vasey SY, Brainsky A. Efficacy of eltrombopag in management of bleeding symptoms associated with chronic immune thrombocytopenia. Blood Coagul Fibrinolysis. 2013 Apr;24(3):284-96. doi: 10.1097/MBC.0b013e32835fac99. PMID 23492914
- [Derived] Saleh MN, Bussel JB, Cheng G, Meyer O, Bailey CK, Arning M, Brainsky A; EXTEND Study Group. Safety and efficacy of eltrombopag for treatment of chronic immune thrombocytopenia: results of the long-term, open-label EXTEND study. Blood. 2013 Jan 17;121(3):537-45. doi: 10.1182/blood-2012-04-425512. Epub 2012 Nov 20. PMID 23169778
- [Derived] Fogarty PF, Tarantino MD, Brainsky A, Signorovitch J, Grotzinger KM. Selective validation of the WHO Bleeding Scale in patients with chronic immune thrombocytopenia. Curr Med Res Opin. 2012 Jan;28(1):79-87. doi: 10.1185/03007995.2011.644849. Epub 2011 Dec 20. PMID 22117897
- [Derived] Signorovitch J, Brainsky A, Grotzinger KM. Validation of the FACIT-fatigue subscale, selected items from FACT-thrombocytopenia, and the SF-36v2 in patients with chronic immune thrombocytopenia. Qual Life Res. 2011 Dec;20(10):1737-44. doi: 10.1007/s11136-011-9912-9. Epub 2011 May 1. PMID 21533818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were previously enrolled in a study of eltrombopag: TRA100773A, TRA100773B, TRA102537/RAISE, or TRA108057/REPEAT. Eligibility of consenting subjects was assessed during the screening period of up to 28 days prior to Day 1 of treatment.
Groups:
- Eltrombopag: Open-label eltrombopag was supplied in 25, 50, 75 mg tablets. All subjects started at 50mg once daily and dose was increased or decreased based on platelet count (target range 50-200Gi/L). Alternate days and interruption of dosing was permitted to maintain target range of platelet count. Doses could range from 25 to 75mg. Subjects could remain on treatment up to 2 years.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 302
Subjects From TRA100773A | 51
Subjects From TRA100773B | 61
Subjects From TRA102537 Raise | 146
Subjects From TRA108057 Repeat | 43
Unknown - Not From Previous Trial | 1 (Mistakenly enrolled (not in any of the 3 trials) On 50 mg/d eltrombopag for 18 days and withdrawn)
Completed | 135
Not Completed | 167
Not completed — Adverse Event | 42
Not completed — Withdrawal by Subject | 39
Not completed — Various -follow up w clinical team | 39
Not completed — Lack of Efficacy | 32
Not completed — Non-compliance | 8
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.9 (15.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 101
Concomitant ITP Medication at Baseline [Number; unit: Participant]
  Yes | 101
  No | 201
Splenectomy Status at Baseline [Number; unit: Participants]
  Yes | 115
  No | 187
Baseline Platelet Count [Number; unit: Participants]
  <30 Gi/L | 211
  30 - 50 Gi/L | 52
  > 50 Gi/L | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of On-Therapy Adverse Events (Safety Population)
Description: All safety evaluation findings considered to be adverse events are reported in the Adverse Event section.
Time Frame: Start date was the first dose of investigational product and up to the day after the last dose . Post-therapy: start date was more than 1 day after the last dose and up to 30 days after last dose of investigational product up to week 364
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  Any adverse event | 277
  Any serious adverse event | 96
  Adverse events related to study medication | 133
  Adverse events leading to withdrawal | 41
  Serious adverse events leading withdrawal | 28

2. Secondary Outcome: Subjects Achieving Maximum Platelet Counts Greater Than or Equal to 30 Gi/L or 50 Gi/L in the Absence of Rescue Medication
Description: Subjects who achieved maximum platelet count at least once during treatment. All platelet counts after an on-study splenectomy are not classed as responses.
  Platelet counts within 7 days after a platelet transfusion are not classed as responses.
  Platelet counts while taking an increased ITP medication or within 6 weeks after the end of an increased ITP medication are not classed as responses.
Time Frame: Baseline up to 2 years
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  Baseline Platelet counts >= 30 Gi/L, | 91
  Baseline Platelet counts >= 50 Gi/L, | 42
  Maximum Platelet Count >= 30 Gi/L | 276
  Maximum Platelet Count >= 50 Gi/L | 259

3. Secondary Outcome: Summary of Subjects Achieving Platelet Count Levels by Week, in the Absence of Rescue Medication
Description: If a subject has more than 1 platelet count result within a week, the lowest value observed is used to determine response. All platelet counts after an on-study splenectomy are not classed as responses. Platelet counts within 7 days after a platelet transfusion are not classed as responses.
  Platelet counts while taking an increased ITP medication or within 6 weeks after the end of an increased ITP medication are not classed as responses.
Time Frame: Baseline up to Year 7/Week 364
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  Baseline Platelet counts >= 30 Gi/L, n=302 | 91
  Baseline Platelet counts >= 50 Gi/L, n=302 | 42
  Week 1 Platelet Count >= 30 Gi/L n=293 | 172
  Week 1 Platelet Count >= 50 Gi/L n=293 | 127
  Week 2 Platelet Count >= 30 Gi/L n=288 | 199
  Week 2 Platelet Count >= 50 Gi/L n=288 | 165
  Week 3 Platelet Count >= 30 Gi/L n=275 | 192
  Week 3 Platelet Count >= 50 Gi/L n=275 | 159
  Week 4 Platelet Count >= 30 Gi/L n=275 | 192
  Week 4 Platelet Count >= 50 Gi/L n=275 | 149
  Week 5 Platelet Count >= 30 Gi/L n=274 | 197
  Week 5 Platelet Count >= 50 Gi/L n=274 | 159
  Week 6 Platelet Count >= 30 Gi/L n=276 | 203
  Week 6 Platelet Count >= 50 Gi/L n=276 | 169
  Week 12 Platelet Count >= 30 Gi/L n=197 | 147
  Week 12 Platelet Count >= 50 Gi/L n=197 | 120
  Month 6/Week 26 Platelet Count >= 30 Gi/L n=130 | 93
  Month 6/Week 26 Platelet Count >= 50 Gi/L n=130 | 82
  Year 1/Week 52 Platelet Count >= 30 Gi/L n=83 | 62
  Year 1/Week 52 Platelet Count >= 50 Gi/L n=83 | 50
  Year 1.5/Week 78 Platelet Count >= 30 Gi/L n=63 | 47
  Year 1.5/Week78 Platelet Count >= 50 Gi/L n=63 | 41
  Year 2/Week 104 Platelet Count >= 30 Gi/L n=59 | 46
  Year 2/Week 104 Platelet Count >= 50 Gi/L n=59 | 42
  Year 2.5/Week 130 Platelet Count >= 30 Gi/L n=42 | 32
  Year 2.5/Week 130 Platelet Count >= 50 Gi/L n=42 | 28
  Year 3/Week 156 Platelet Count >= 30 Gi/L n=27 | 22
  Year 3/Week 156 Platelet Count >= 50 Gi/L n=27 | 19
  Year 3.5/Week 182 Platelet Count >= 30 Gi/L n=23 | 19
  Year 3.5/Week 182 Platelet Count >= 50 Gi/L n=23 | 17
  Year 4/Week 208 Platelet Count >= 30 Gi/L n=17 | 12
  Year 4/Week 208 Platelet Count >= 50 Gi/L n=17 | 11
  Year 4.5/Week 234 Platelet Count >= 30 Gi/L n=15 | 13
  Year 4.5/Week 234 Platelet Count >= 50 Gi/L n=15 | 12
  Year 5/Week 260 Platelet Count >= 30 Gi/L n=9 | 6
  Year 5/Week 260 Platelet Count >= 50 Gi/L n=9 | 6
  Year 5.5/Week 286 Platelet Count >= 30 Gi/L n=9 | 7
  Year 5.5/Week 286 Platelet Count >= 50 Gi/L n=9 | 7
  Year 6/Week 312 Platelet Count >= 30 Gi/L n=9 | 7
  Year 6/Week 312 Platelet Count >= 50 Gi/L n=9 | 7
  Year 6.5/Week 338 Platelet Count >= 30 Gi/L n=5 | 3
  Year 6.5/Week 338 Platelet Count >= 50 Gi/L n=5 | 3
  Year 7/Week 364 Platelet Count >= 30 Gi/L n=3 | 3
  Year 7/Week 364 Platelet Count >= 50 Gi/L n=3 | 3

4. Secondary Outcome: Number of Subjects Who Responded to Eltrombopag in a Previous Study and Who Respond to Retreatment With a Rise in Platelet Count to Either ≥ 50,000/µL or ≥30,000/µL
Description: Responder in TRA100773: Platelet count 50 Gi/L and 2 x baseline (BL) at last on-treatment assessment. Responders in EXTEND: Platelet count 50 Gi/L and 2 x baseline (BL), 50 Gi/L, and 30 Gi/L at any time. Responder in RAISE: Platelet count 50GI/L and 2 x baseline at Week 6 assessment. Responders in EXTEND: Platelet count 50 Gi/L and 2 x baseline, 50 Gi/L, and 30 Gi/L at any time. Responder in REPEAT: Platelet count 50 GI/L and 2 x baseline (BL) at Week 6 assessment in Cycle 1. Responders in EXTEND: Platelet count 50 Gi/L and 2 x baseline (BL) 50 Gi/L, and 30 Gi/L at any time.
Time Frame: Baseline up to 2 years
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  TRA100773 Responders >= 50 Gi/L in EXTEND, n=51 | 49
  TRA100773 >=50 Gi/L and 2 x BL in EXTEND, n=51 | 47
  TRA100773 Responders >= 30 Gi/L in EXTEND, n=51 | 49
  RAISE Responders >= 50 Gi/L in EXTEND, n=59 | 54
  RAISE >= 50 Gi/L and 2 x BL in EXTEND, n=59 | 53
  RAISE Responders >= 30 Gi/L in EXTEND, n=51 | 55
  REPEAT Responders >= 50 Gi/L in EXTEND, n=36 | 33
  REPEAT>= 50 Gi/L and 2 x BL in EXTEND, n=36 | 33
  REPEAT Responders >= 30 Gi/L in EXTEND, n=36 | 35

5. Secondary Outcome: Number of Participants With Reduction and/or Sparing of Concomitant ITP Therapies, While Maintaining a Platelet Count ≥ 50,000/mL.
Description: Sustain reduct: Sustained reduction 1 Denominator is number of subjects taking an ITP medication at baseline. 2 Denominator is number of subjects with a sustained reduction. Note: Sustained reduction defined as reduction from baseline in dose and/or frequency which is maintained for at least 4 weeks. Excludes sustained reductions started more than 1 day after last dose.
Time Frame: Baseline up to 2 years
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  ITP medication at baseline | 101
  Sustain reduct or stop at least 1 med [1] n=101 | 71
  Permanently stopping at least 1 ITP med [1] n=101 | 53
  Sustained reduction[1] n=101 | 70
  Maximum sustained reduction ≥ 24 weeks[2] n=70 | 66

6. Secondary Outcome: Number of Subjects Who Required Rescue Therapy During Treatment With Eltrombopag.
Description: Rescue treatment is defined as a composite of: new ITP medication, increased dose of a concomitant ITP medication, platelet transfusion, and splenectomy. Subjects may have received more than 1 type of rescue therapy
Time Frame: Baseline up to 2 years
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  New ITP medication, n=103 | 82
  Increase in dose of ITP med from baseline, n=103 | 27
  Platelet transfusion, n=103 | 21
  Splenectomy, n=103 | 3

7. Secondary Outcome: Maximum ITP Bleeding Score at Any Time During the Study During All Stages.
Description: The ITP bleeding score is a tool which has been designed specifically to assess the bruising and bleeding in patients with ITP across body sites, ranging from mild to severe. The WHO Grades were dichotomized into the following categories: - Grade 0, No bleeding -Grade 1 to 4, Any bleeding -Grade 0 to 1: No clinically significant bleeding -Grade 2 to 4 Clinically significant bleeding
Time Frame: Baseline up to 2 years
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 302
Participants
  Epistaxis n=300 Grade 0 | 204
  Epistaxis n=300 Grade 1 | 65
  Epistaxis n=300 Grade 2 | 31
  Gastrointestinal n=300 Grade 0 | 264
  Gastrointestinal n=300 Grade 1 | 26
  Gastrointestinal n=300 Grade 2 | 10
  Genitourinary n=300 Grade 0 | 262
  Genitourinary n=300 Grade 1 | 29
  Genitourinary n=300 Grade 2 | 9
  Gynecologic n=108 Grade 0 | 68
  Gynecologic n=108 Grade 1 | 15
  Gynecologic n=108 Grade 2 | 25
  Intracerebral hemorrhage n=300 Grade 0 | 297
  Intracerebral hemorrhage n=300 Grade 1 | 3
  Intracerebral hemorrhage n=300 Grade 2 | 0
  Ocular n=300 Grade 0 | 258
  Ocular n=300 Grade 1 | 37
  Ocular n=300 Grade 2 | 5
  Oral n=300 Grade 0 | 191
  Oral n=300 Grade 1 | 81
  Oral n=300 Grade 2 | 28
  Pulmonary n=300 Grade 0 | 287
  Pulmonary n=300 Grade 1 | 13
  Pulmonary n=300 Grade 2 | 0
  Skin, ecchymosis n=300 Grade 0 | 74
  Skin, ecchymosis n=300 Grade 1 | 159
  Skin, ecchymosis n=300 Grade 2 | 67
  Skin, petechiae n=300 Grade 0 | 142
  Skin, petechiae n=300 Grade 1 | 126
  Skin, petechiae n=300 Grade 2 | 32

8. Secondary Outcome: Best Post-Baseline Change in SF-36v2 Questionnaire Score From Any Time Point Compared With Baseline
Description: The SF-36v2 assessment tool was used to obtain information about subjects' general health status and health-related quality of life. Until a formal assessment of minimal clinically important differences (MCID) is performed, changes from baseline of more than 0.5 standard deviations are suggested as clinically meaningful. Scores were transformed to a 0-100 point scale, with higher scores representing more positive answers. Scores were normalized to have a mean of 50 and SD of 10 to allow for comparison with outcomes from other chronic diseases. Recall period is the past week prior to administration. The change in scores was measured at the transitioning period and immediately prior to withdrawal/completion over 2 years, and the mean of these measurements was recorded to calculate the change from baseline and the best post baseline change score was reported for the entire group
Time Frame: Baseline, beginning of each stage, change in therapy and minimum frequency of every 3 months during stages, prior to early discontinuation, up to 2 years
Measure: Mean (95% Confidence Interval); unit: Points on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 290
Points on a scale
  SF-36v2 Physical function (n=273 | 12.0 [9.6 to 14.5]
  SF-36v2 Physical role (n=273) | 14.2 [11.5 to 16.9]
  SF-36v2 Bodily pain (n=273) | 14.5 [11.6 to 17.4]
  SF-36v2 General health (n=273) | 11.1 [9.0 to 13.1]
  SF-36v2 Vitality (n=290) | 13.9 [11.6 to 16.3]
  SF-36v2 Social function (n=290) | 12.6 [10.2 to 15.1]
  SF-36v2 Emotional role (n=290) | 11.4 [8.7 to 14.0]
  SF-36v2 Mental health (n=290) | 11.3 [9.4 to 13.3]
  SF-36v2 Physical component summary (n=273) | 5.3 [4.5 to 6.2]
  SF-36v2 Mental component summary (n=290) | 5.8 [4.6 to 6.9]

9. Secondary Outcome: Best Post-Baseline Change in the Short Form of the Motivation and Energy Scale (MEI-SF) From Any Time Point Compared With Baseline
Description: The MEI-SF (18 questions) was used to measure the reductions in mental energy, physical energy, and social motivation, either as symptoms of chronic ITP or as a side effect of pharmacotherapy. Minimal clinically important differences are estimated as 0.5 standard deviations or 7.5 points. All items use either a 7-level (0 to 6) or 5-level (0 to 4) response scale; items with a 5-level response scale were rescaled to 7-levels, and items were reverse-scored as necessary such that higher scores represent higher HRQoL Total score ranges from 0 to 108 points. Recall period is past week prior to administration. The change in scores was measured at the transitioning period and immediately prior to withdrawal/completion over 2 years, and the mean of these measurements was recorded to calculate the change from baseline and the best post baseline change score was reported for the entire group
Time Frame: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Points on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 292
Points on a scale | 11.3 [9.1 to 13.5]

10. Secondary Outcome: Best Post-Baseline Change in the FACIT-Fatigue 13 Item Subscale Score From Any Time Point Compared to Baseline
Description: The FACIT-Fatigue consists of 13 questions in which patients rate the frequency (0-4) of symptoms of fatigue, in terms of tiredness, weakness, and fatigue Items were reverse-scored as necessary such that higher scores represent higher HRQoL Total score ranges from 0 to 52.Using anchor-based estimates, the minimally important difference in this subscale is 3.0 points.
  Recall period is past week prior to administration. The change in scores was measured at the transitioning period and immediately prior to withdrawal/completion over 2 years, and the mean of these measurements was recorded to calculate the change from baseline and the best post baseline change score was reported for the entire group
Time Frame: as for outcome 8
Population: ITT
Measure: Mean (95% Confidence Interval); unit: Points on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 291
Points on a scale | 6.9 [5.7 to 8.1]

11. Secondary Outcome: Best Post-Baseline Change in the FACT-TH6 at Any Time Point Compared to Baseline
Description: The FACT-TH6 consists of 6 questions in which patients rate (0-4) their general degree of worry related to bleeding and bruising, and resulting activity impairment and frustration. Although the six items do not constitute a formal domain or subscale of the FACT-Th assessment tool, these items had been identified by focus groups of patients with chronic ITP as important indicators of their HRQoL. Items were reverse-scored as necessary such that higher scores represent higher HRQoL. Total scores ranged from 0 to 24. Recall period is not specified. The change in scores was measured at the transitioning period and immediately prior to withdrawal/completion over 2 years, and the mean of these measurements was recorded to calculate the change from baseline and the best post baseline change score was reported for the entire group
Time Frame: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Points on a scale
Arm/Group | Eltrombopag
Number analyzed (Participants) | 288
Points on a scale | 4.0 [3.4 to 4.6]

ADVERSE EVENTS:
Time Frame: Treatment + 1 Day: start date was between the first dose of investigational product and up to the day after the last dose . Post-therapy: start date was more than 1 day after the last dose and up to 30 days after last dose of investigational product
Groups:
- Eltrombopag, Treatment + 1 Day: Eltrombopag, Treatment + 1 day
- Eltrombopag, >1 to 30 Days Post-Therapy: Eltrombopag, >1 to 30 Days Post-Therapy
Arm/Group | Eltrombopag, Treatment + 1 Day | Eltrombopag, >1 to 30 Days Post-Therapy
Serious Adverse Events (participants affected / at risk) | 96/302 | 10/302
Other Adverse Events (participants affected / at risk) | 253/302 | 28/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag, Treatment + 1 Day (N=302) | Eltrombopag, >1 to 30 Days Post-Therapy (N=302)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Bone marrow oedema (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Splenic cyst (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 16 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Choroidal neovascularisation (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Medical device pain (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Wound infection (Infections and infestations) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 4 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 3 | 0
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Toxic neuropathy (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag, Treatment + 1 Day (N=302) | Eltrombopag, >1 to 30 Days Post-Therapy (N=302)
Anaemia (Blood and lymphatic system disorders) | 26 | 1
Abdominal pain (Gastrointestinal disorders) | 18 | 0
Abdominal pain upper (Gastrointestinal disorders) | 18 | 1
Constipation (Gastrointestinal disorders) | 26 | 2
Diarrhoea (Gastrointestinal disorders) | 46 | 3
Nausea (Gastrointestinal disorders) | 34 | 1
Vomiting (Gastrointestinal disorders) | 19 | 2
Fatigue (General disorders) | 50 | 4
Influenza like illness (General disorders) | 25 | 1
Pyrexia (General disorders) | 27 | 2
Bronchitis (Infections and infestations) | 25 | 0
Cystitis (Infections and infestations) | 16 | 0
Influenza (Infections and infestations) | 29 | 0
Nasopharyngitis (Infections and infestations) | 74 | 2
Pharyngitis (Infections and infestations) | 21 | 0
Sinusitis (Infections and infestations) | 20 | 1
Upper respiratory tract infection (Infections and infestations) | 69 | 5
Urinary tract infection (Infections and infestations) | 32 | 2
Viral infection (Infections and infestations) | 23 | 0
Alanine aminotransferase increased (Investigations) | 23 | 0
Aspartate aminotransferase increased (Investigations) | 21 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 0
Dizziness (Nervous system disorders) | 26 | 0
Headache (Nervous system disorders) | 86 | 3
Insomnia (Psychiatric disorders) | 27 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 1
Rash (Skin and subcutaneous tissue disorders) | 25 | 0
Hypertension (Vascular disorders) | 22 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.